CLINICAL TRIAL: NCT06244095
Title: Comparative Effects of Perturbation and Trunk Control Training in Children With Cerebral Palsy
Brief Title: Effects of Perturbation Therapy and Trunk Control Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0737
Record Dates: First submitted 2023-12-25; First posted 2024-02-06 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Perturbation Therapy; Trunk control training.
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perturbation Therapy (Experimental): Perturbation Therapy will be given to this group.
  Interventions: Other: Perturbation Therapy
- Trunk Control Therapy (Active Comparator): Trunk control activities will be given to this group.
  Interventions: Other: Trunk Control Therapy

INTERVENTIONS:
Other: Perturbation Therapy — The applicants were instructed to perform various exercises, including rotating their trunks, tossing a ball, and maintaining pelvis neutrality. They were also asked to reach the toy sideways with one hand. The 6-week intervention was conducted four days a week for 60 minutes each day, focusing on trunk rotation, standing, tossing, and catching the ball in various directions. The training sessions lasted for 20 minutes each.
  Arms: Perturbation Therapy
Other: Trunk Control Therapy — For the duration of each session, the manual pushes and pulls were administered around once per minute and lasted for 20 minutes. A platform that can be moved in four directions.Choosing to step and stroll when there is an outside disturbance. When routine motions such as sit-to-stand transitions, disruptions are applied when standing, walking, or other activities. Training with continuous disruptions simulates scenarios such as uneven terrain. Both rope and cable excursions are above ground and last for 20 minutes. Briefly explain the platform to the participants. Asked the participants to push the torso and waist against the wall during the session. Emerging barriers during training sessions like small obstacles (e.g. pair of bricks) then Lean the participants with the support of the therapist and let them go. Asked them to Step on a mushy or slick surface in session for 20 minutes. Each intervention session took place for 60 minutes per day four days of week for 6 weeks.
  Arms: Trunk Control Therapy

SUMMARY:
A postural perturbation refers to unexpected change in conditions that upsets the body's harmony and displaces its posture. These perturbations can be sensory in nature, such as vestibular perturbations resulting from electrical stimulation, visual perturbations caused by a moving room or graphical images, or somatosensory perturbations caused by muscle vibrations. The body's reactions to these sensory perturbations may be based on the perception of instability rather than actual imbalance. Trunk control plays a vital role in various aspects of daily life, including balance, walking, and overall functional abilities. Children with cerebral palsy (CP), who experience limitations in their ability to move, often expend more energy compared to their healthy peers.

DETAILED DESCRIPTION:
This study will be randomized clinical trial used to compare the effects of Perturbation and trunk control training in children with Cerebral Palsy. Subjects meeting the predetermined inclusion and exclusion criteria will be divided into two groups using lottery method. Pre-assessment will be done using Berg balance scale, functional Independent measures and TUG test as objective measurements. Subjects in one group will be treated using Perturbation therapy and the other one will be treated with Trunk control training. Both groups had three treatment sessions per week, for 4 weeks, and the total time for every session was about 30-45 minutes. A postural perturbation refers to unexpected change in conditions that upsets the body's harmony and displaces its posture. These perturbations can be sensory in nature, such as vestibular perturbations resulting from electrical stimulation, visual perturbations caused by a moving room or graphical images, or somatosensory perturbations caused by muscle vibrations. The body's reactions to these sensory perturbations may be based on the perception of instability rather than actual imbalance. On the other hand, "mechanical perturbations" physically displace the body segments, potentially leading to a shift in the overall center of mass or actual imbalance. Even small displacements of a single body segment, like the head, can elicit minor muscle responses throughout the body

ELIGIBILITY:
Inclusion Criteria:

* Kids that suffer from cerebral palsy.
* Ages span from 5 to 10 years.
* Both males and females were represented.
* During the preceding half-year, there was no orthopedic surgery or spasticity-reduction intervention.
* No significant lower limb muscular contraction

Exclusion Criteria:

* Individuals suffering from sensory, proprioceptive, cognitive, and perceptual impairments, as well as those with contractures.
* Any neurological disease that impairs balance, including orthopedic disorders
* Individual experiencing seizures and has undergone any prior surgical treatments.
* Uncorrected visual issues

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Pediatric Berg balance scale (PBBS) | 6weeks
  BBS is 14 Item rating 5-point ordinal Scale, used to evaluate the balance in elderly population and other neurological conditions. It is easy to administer and doesn't require specialized training and takes 15- 20 mins. The maximum scoring in BBS is 56.
Functional Independent Measures (FIM | 6weeks
  The Functional Independence Measure (FIM) provides a seven level ordinal scale for measuring functional performance on 18 activities considered essential for daily living. In routine practice, the scores on the individual activities are usually summed giving a total FIM score that ranges from 18 to 126.
Timed Up and Go Test (TUGT) | 6weeks
  It is prognostic test to assess mobility and to identify the individuals with a risk of fall. TUG is time performance of getting up from chair, walking 3 m, turning around and walking back to sit down again. Timed Up and Go test is recommended by American Geriatrics Society, British Geriatric Society for screening risk of falls. An older who takes more than 12 seconds to complete the TUG is at the highest risk for falling

CONTACTS AND LOCATIONS:
Overall Officials: Zirwa Afzal, MS*, Principal Investigator — Riphah International University
Locations (1):
- Imran Amjad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horak FB, Earhart GM, Dietz V. Postural responses to combinations of head and body displacements: vestibular-somatosensory interactions. Exp Brain Res. 2001 Dec;141(3):410-4. doi: 10.1007/s00221-001-0915-6. PMID 11715086